CLINICAL TRIAL: NCT06565195
Title: A Randomized, Double-blind (Sponsor-unblinded), Placebo-controlled, Single-ascending-dose Study in Healthy Volunteers and a Double-blind (Sponsor-unblinded), Placebo-controlled, Multiple-ascending-dose Study in Patients With Parkinson's Disease to Evaluate the Safety, Tolerability, and PK/PD of LY3962681
Brief Title: A Clinical Trial of LY3962681 in Healthy Volunteers and in Patients With Parkinson's Disease
Acronym: PROSPECT-PD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Prevail Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: J5F-MC-OOAA
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Healthy volunteers
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both the SAD and MAD studies are double blinded (sponsor unblinded); that is, both the participants and the site personnel are blinded to the study intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3962681 (SAD) (Experimental): Single ascending dose of LY3962681 or placebo (aCSF) administered intrathecally (IT) to healthy volunteers.
  Interventions: Drug: LY3962681; Other: Placebo (aCSF)
- LY3962681 (MAD) (Experimental): Multiple ascending doses of LY3962681 or placebo (aCSF) administered IT to participants with Parkinson's disease.
  Interventions: Drug: LY3962681; Other: Placebo (aCSF)

INTERVENTIONS:
Drug: LY3962681 — IT injection
Other: Placebo (aCSF) — IT injection

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and PK/PD of LY3962681 in healthy volunteers and patients with Parkinson's disease.

The study will be comprised of two parts, the Single Ascending Dose (SAD) study and the Multiple Ascending Doses (MAD) study. During the SAD portion of the study, healthy volunteers will receive a single dose of LY3962681 or placebo (artificial cerebrospinal fluid (aCSF), no active drug) given into the spinal fluid. During the MAD portion of the study, patients with Parkinson's disease will receive two doses of either LY3962681 or placebo (aCSF) administered into the spinal fluid.

* The treatment period in the SAD study will be 1 day. The treatment period in the MAD study will be 2 days, 12 to 24 weeks apart.
* The follow-up period in the SAD study will be up to 52 weeks. The follow-up period in the MAD study will be up to 52 weeks post Dose 2.

ELIGIBILITY:
Inclusion Criteria:

* Participant is overtly healthy as determined by medical evaluation. Rescreening is allowed in this study.
* A Montreal Cognitive Assessment score greater than or equal to 24.
* Stable use of background medications at least 8 weeks prior to IP administration, including but not limited to those used for treatment of Parkinson's disease (including deep brain stimulation), and the investigator must expect that participant can tolerate a minimum of 6 months without dose adjustment.

MAD study only

* Participant has a diagnosis of Parkinson's disease per UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria.
* Modified Hoehn and Yahr Stage 1 to 2.5 in the practically defined OFF state.
* A positive result on CSF alpha-synuclein Seed Amplification Assay. (A prior positive result [within 1 year of screening] accepted with sponsor approval if patient did not participate in another Parkinson's disease clinical trial during this period.) (US and Japan only)
* UPSIT score of 10 percentile or less, corrected for age and sex (EU and UK only).
* An abnormal DaT-SPECT consistent with parkinsonism. (History of an abnormal DaTSPECT with the report confirmed by study investigator will be accepted.)
* For participants not taking Parkinson's disease medications, not expected to initiate treatment within 6 months.
* Have a body weight within 40 kg (88 pounds) to 110 kg (242 pounds), inclusive, and body mass index within the range of 17 to 34 kg/m^2, inclusive.

Exclusion Criteria:

* MAD study only: Significant neurological disease affecting the central nervous system other than Parkinson's disease that may be a cause for the participant's clinical symptoms or may confound study objectives.
* Current concomitant disease or serious or unstable illnesses, including central nervous system (SAD study only), cardiovascular, hepatic, renal, gastroenterology, respiratory, endocrinologic, neurologic (MAD study only: other than Parkinson's disease), psychiatric, immunologic, or hematologic disease and other conditions that, in the investigator's opinion, could interfere with the conduct of the study or that would, in the opinion of the investigator, pose an unacceptable safety risk to the participant.
* Participant is generally frail or has any medical disorders that, in the opinion of the investigator, could interfere with study-related procedures (including safe performance of IT injection or LP), such as prohibitive spinal diseases, bleeding diathesis, clinically significant coagulopathy, thrombocytopenia, or increased intracranial pressure.
* Have a 12-lead ECG abnormality at screening that, in the opinion of the investigator, increases the risks associated with participating in the study or may confound ECG data analysis.
* MAD study only: Treatment with continuous intestinal delivery Parkinson's disease medication (for example, Duodopa).

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2029-05-05 (Estimated); Study Completion 2029-05-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events (SAEs) | Up to 76 weeks
Incidence of Treatment Emergent Adverse Events (TEAEs) | Up to 76 weeks
Number of discontinuations due to Adverse Events (AEs) | Up to 76 weeks

SECONDARY OUTCOMES:
LY3962681 Maximum Observed Concentration (Cmax) | Up to 76 weeks
LY3962681 area under the concentration versus time curve | Up to 76 weeks
Change from baseline in CSF total alpha-synuclein | Up to 76 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Travis Lewis, Study Director — Prevail Therapeutics, a Wholly Owned Subsidiary of Eli Lilly and Company
Locations (4):
- Austin Clinic PPD, Austin, Texas, United States
- Japan (3):
  - Ehime University Hospital, Tōon, Ehime
  - Oita University Hospital, Yufu, Oita Prefecture
  - P-One Clinic, Keikokai Medical Corporation, Hachiōji, Tokyo

IPD SHARING:
Plan to Share IPD: No